CLINICAL TRIAL: NCT05540028
Title: A Phase 1, Multicenter, Randomized, Active-Controlled, Observer-Blind, Study to Evaluate the Safety, Tolerability, and Immunogenicity of Inventprise's 25-Valent Pneumococcal Conjugate Vaccine in Healthy PCV-Naïve Adults (18 Through 40 Years)
Brief Title: Study to Evaluate a 25-Valent Pneumococcal Conjugate Vaccine
Acronym: IVT PCV-25
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inventprise Inc. (Industry)
Collaborators: Canadian Center for Vaccinology (Other); Vaccine Evaluation Center, Canada (Other); PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA 096
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Pneumococcal Vaccines

STUDY DESIGN:
Intervention Model Description: Single center, randomized, active-controlled, observer-blind Phase 1study in which adults were randomized in a 1:1 ratio to evaluate safety and tolerability of IVT PCV 25 to comparator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult Cohort Group 1 (Experimental): Participants will receive a single 0.5mL dose of IVT PCV-25 administered by intramuscular injection on Day 1
  Interventions: Biological: IVT PCV-25
- Adult Cohort Group 2 (Active Comparator): Participants will receive a single 0.5mL dose of PCV 20 administered by intramuscular injection on Day 1
  Interventions: Biological: PCV 20

INTERVENTIONS:
Biological: IVT PCV-25 — 25 valent pneumococcal conjugate vaccine
  Arms: Adult Cohort Group 1
Biological: PCV 20 — 20 valent pneumococcal conjugate vaccine
  Arms: Adult Cohort Group 2

SUMMARY:
A first-in-human, Phase 1 trial to evaluate safety, tolerability, and immunogenicity of Inventprise's (IVT) 25-valent pneumococcal conjugate vaccine (IVT PCV-25)

DETAILED DESCRIPTION:
A first-in-human, multicenter, randomized, active-controlled, observer-blind Phase 1 study of IVT PCV-25 designed to evaluate the safety, tolerability, and immunogenicity of the vaccine. Adult subjects will be randomized 1:1 to receive either IVT PCV-25 or Prevnar 20™.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are 18 through 40 years old on the day of randomization (Day 1).
* Subject, or subject's LAR, must provide voluntary written informed consent for the subject to participate in the study.
* Subject or subject's LAR must be able to comprehend and comply with study requirements and procedures and must be willing and able to return for all scheduled follow-up visits.
* There will be an allowance though not a requirement for COVID-19 vaccination in all participants in compliance with Canadian national recommendations.
* Adult female subjects who are not surgically sterile must have a negative serum pregnancy test at screening and negative urine pregnancy test prior to vaccination.

Exclusion Criteria:

* Use of any investigational medicinal product within 90 days prior to randomization or planned use of such a product during the period of study participation.
* Adults who have previously been vaccinated against S. pneumoniae.
* History of microbiologically confirmed invasive disease caused by S. pneumoniae.
* History of allergic disease or history of a serious reaction to any prior vaccination or known hypersensitivity to any component of the study vaccines.
* Known or suspected allergy to PEG.
* History of angioedema.
* Any abnormal vital sign deemed clinically relevant by the PI.
* Acute illness (moderate or severe) and/or fever (body temperature of ≥ 38.0°C)
* Use of antibiotics (oral or parenteral) within 5 days of randomization.
* History of administration of any non-study vaccine (e.g. influenza; COVID-19 vaccine) within 14 days of first administration of study vaccine or planned vaccination prior to 14 days post-vaccination blood draw.
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressant or other immune modifying drugs prior to the administration of the study vaccine (and within the 6 months prior to administration of the study vaccine in the case of adults), including the use of glucocorticoids. The use of topical and inhaled glucocorticoids will be permitted.
* Administration of immunoglobulins and/or any blood products within the 6 months prior to administration of the study vaccine, or anticipation of such administration during the study period.
* History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding (e.g., thalassemia, coagulation factor deficiencies, severe anemia).
* Any medical or social condition that in the opinion of the PI , may interfere with the study objectives, pose a risk to the subject, or prevent the subject from completing the study follow-up.
* Subject is an employee of, or direct descendant (child or grandchild) of any person employed by the Sponsor, PATH, the CRO, the PI.
* Any screening laboratory test result outside the normal range and with toxicity score ≥ 2, unless allowed by the PI and PATH Medical Officer when a toxicity score and the normal range overlap significantly. A subject may repeat each laboratory assessment once during the screening period, with the most recent laboratory value being used for evaluation of exclusion criteria.
* A positive serologic test for human immunodeficiency virus (HIV)-1 or HIV-2 (HIV 1/2 Ab), hepatitis B (HBsAg) or hepatitis C (HCV Ab).
* History of malignancy, excluding non-melanoma skin and cervical carcinoma in situ.
* Recent history (within the past year) or signs of alcohol or substance abuse.
* History of major psychiatric disorder.
* Female adult subjects who are pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Adult Safety: solicited local and systemic adverse events | 7 days post-vaccination (Day 8)
  Number and severity of solicited local and systemic adverse events (AEs)
Adult Safety: clinically significant hematological and biochemical measurements | 7 days post-vaccination (Day 8)
  Number, severity, and relatedness of clinically significant hematological and biochemical measurements
Adult Safety: unsolicited adverse events | 28 days post-vaccination (Day 29)
  Number, severity, and relatedness of all unsolicited AEs
Adult Safety: related serious adverse events | through 6 months post last vaccination (Day 169)
  Number, severity, and relatedness of serious adverse events (SAEs)
Adult Safety: newly diagnosed chronic medical conditions | through 6 months post last vaccination (Day 169)
  Number of newly diagnosed chronic medical conditions

SECONDARY OUTCOMES:
Adult Immunogenicity: immunoglobulin G (IgG) geometric mean concentration (GMC) | 28 days post-vaccination (Day 29)
  Serotype-specific IgG GMCs
Adult Immunogenicity: Geometric Mean Fold Rise (GMFR) | 28 days post-vaccination (Day 29)
  Geometric Mean Fold Rise (GMFR) from baseline in serotype-specific IgG GMCs
Adult Immunogenicity: opsonophagocytosis assay (OPA) geometric mean titers (GMTs) | 28 days post-vaccination (Day 29)
  Serotype-specific OPA GMTs
Adult Immunogenicity: GMFR OPA GMTs | 28 days post-vaccination (Day 29)
  GMFR (from baseline) in serotype-specific OPA GMTs

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Langley, MD, MSc, FRCPC, Principal Investigator — Canadian Center for Vaccinology
Locations (1):
- Canadian Center for Vaccinology, IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Plan to be defined at a later date
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Plan to be defined at a later date
Access Criteria: Plan to be defined at a later date

REFERENCES:
- [Derived] Langley JM, Sadarangani M, Ockenhouse C, Barreto L, Ye L, Tang Y, Breeze JL, Feser J, Hosken NA, Andi-Lolo I, Tasker SA, Halperin SA; Canadian Immunization Research Network. Safety and immunogenicity of a 25-valent pneumococcal conjugate vaccine in pneumococcal vaccine-naive healthy adults: Results from 2 randomised, controlled clinical trials. Vaccine. 2026 Jan 22;75:128236. doi: 10.1016/j.vaccine.2026.128236. Online ahead of print. PMID 41576705